CLINICAL TRIAL: NCT01426607
Title: VASO-AM :Impact of Oral Appliance Therapy on Endothelial Function in Obstructive Sleep Apnea
Acronym: VASO-AM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PHRC 2010-06
Record Dates: First submitted 2011-06-28; First posted 2011-08-31 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2011-08

CONDITIONS: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AMO (Experimental): Adjustable mandibular repositioning appliance
  Interventions: Device: AMO
- placebo (Placebo Comparator): placebo device in upper jaw
  Interventions: Device: AMO

INTERVENTIONS:
Device: AMO

SUMMARY:
This is a randomized controlled study evaluating the impact of 2 months of oral appliance therapy on endothelial function in patients with severe obstructive sleep apnea syndrome intolerant to continuous positive airway pressure (CPAP) therapy.

ELIGIBILITY:
Inclusion Criteria:

* AHI > 30
* Intolerance to CPAP therapy
* Signed informed consent

Exclusion Criteria:

* Epworth sleepiness scale > 16/24
* Severe cardiac and/or respiratory disease
* BMI>32 kg/m2
* Dental contraindication to oral appliance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
change from baseline to 2-months in reactive hyperemia index (RHI), a validated measurement of endothelial function. | 2 months

SECONDARY OUTCOMES:
change from baseline to 2-months in markers of OSA severity | 2 months
change from baseline to 2-months in blood pressure | 2 months
change from baseline to 2-months in symptoms of OSA | 2 months
evaluate treatment compliance objectively measured by an embedded micro sensor | 15 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU Grenoble, Grenoble
  - CH Le Mans, Le Mans
  - Hopital Saint Antoine, Paris
  - CHU Poitiers, Poitiers

REFERENCES:
- [Derived] Recoquillon S, Pepin JL, Vielle B, Andriantsitohaina R, Bironneau V, Chouet-Girard F, Fleury B, Goupil F, Launois S, Martinez MC, Meslier N, Nguyen XL, Paris A, Priou P, Tamisier R, Trzepizur W, Gagnadoux F. Effect of mandibular advancement therapy on inflammatory and metabolic biomarkers in patients with severe obstructive sleep apnoea: a randomised controlled trial. Thorax. 2019 May;74(5):496-499. doi: 10.1136/thoraxjnl-2018-212609. Epub 2018 Oct 26. PMID 30366971
- [Derived] Gagnadoux F, Pepin JL, Vielle B, Bironneau V, Chouet-Girard F, Launois S, Meslier N, Meurice JC, Nguyen XL, Paris A, Priou P, Tamisier R, Trzepizur W, Goupil F, Fleury B. Impact of Mandibular Advancement Therapy on Endothelial Function in Severe Obstructive Sleep Apnea. Am J Respir Crit Care Med. 2017 May 1;195(9):1244-1252. doi: 10.1164/rccm.201609-1817OC. PMID 28128967